CLINICAL TRIAL: NCT04475991
Title: Phase2, Randomized, Controlled Study to Evaluate the Efficacy and Safety of Maraviroc and/or Favipiravir Plus Standard Therapy in Adult Patients With Severe Non-critical COVID-19"
Brief Title: Safety and Efficacy of Maraviroc and/or Favipiravir With Standard Therapy in Severe COVID-19 Adults
Acronym: COMVIVIR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No more patients complying the selection criteria were available for recruitment
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Collaborators: CCINSHAE. Secretaría de Salud. México (Unknown); Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other); Centro de Investigación en. Enfermedades Infecciosas, Mexico (Other Government)
Responsible Party: Principal Investigator, María Luisa Hernández-Medel, Researcher, Hospital General de México Dr. Eduardo Liceaga
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DI/20/407/04/38
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: COVID-19; CCR5; Cytokine storm; Maraviroc; Favipiravir; RdRP inhibitors
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — Maraviroc; favipiravir

STUDY DESIGN:
Intervention Model Description: 100 participants will be included and allocated in 4 groups of 25 each [Currently used therapy (CT), Maraviroc+CT, Favipiravir+CT and Maraviroc+Favipiravir+CT]. Subjects will be randomized using EPIDAT 4.2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Currently used therapy (CT) only (Active Comparator): Treatment currently used at Hospital General de México "Dr. Eduardo Liceaga" for non-critical COVID patients: Enoxaparin, dexamethasone, and antibiotics if associated bacteremia is present.
  Interventions: Procedure: Curently used therapy for COVID-19 non-critical patients
- Maraviroc+CT (Experimental): Maraviroc AND treatment currently used at Hospital General de México "Dr. Eduardo Liceaga" for non-critical COVID patients.
  Interventions: Drug: Maraviroc + Currently used therapy
- Favipiravir+CT (Experimental): Favipiravir AND treatment currently used at Hospital General de México "Dr. Eduardo Liceaga" for non-critical COVID patients.
  Interventions: Drug: Favipiravir + Currently used therapy
- Maraviroc+Favipiravir+CT (Experimental): Maraviroc AND Favipiravir AND treatment currently used at Hospital General de México "Dr. Eduardo Liceaga" for non-critical COVID patients
  Interventions: Drug: Maraviroc+Favipiravir+CT

INTERVENTIONS:
Drug: Maraviroc + Currently used therapy — Maraviroc tablets. 300 mg bid, given orally for a 10 day period AND CT (Enoxaparin, dexamethasone, and antibiotics if associated bacteremia is present, as per currently used at Hospital General de México "Dr. Eduardo Liceaga")
  Other Names: MVC+CT
  Arms: Maraviroc+CT
Procedure: Curently used therapy for COVID-19 non-critical patients — Enoxaparin, dexamethasone, and antibiotics if associated bacteremia is present, as per currently used at Hospital General de México "Dr. Eduardo Liceaga"
  Other Names: CT only
  Arms: Currently used therapy (CT) only
Drug: Favipiravir + Currently used therapy — Favipiravir tablets 200 mg. given orally for a 7 day period. 1600 mg bid on day 1 and 600 mg tid days 2-7 AND CT (Enoxaparin, dexamethasone, and antibiotics if associated bacteremia is present, as per currently used at Hospital General de México "Dr. Eduardo Liceaga").
  Other Names: FPV+CT
  Arms: Favipiravir+CT
Drug: Maraviroc+Favipiravir+CT — Maraviroc tablets. 300 mg bid, given orally for a 10 day period AND Favipiravir tablets 200 mg. given orally for the first 7 days. 1600 mg bid on day 1 and 600 mg tid days 2-7 AND CT (Enoxaparin, dexamethasone, and antibiotics if associated bacteremia is present, as per currently used at Hospital General de México "Dr. Eduardo Liceaga"")
  Other Names: MVC+FPV+CT
  Arms: Maraviroc+Favipiravir+CT

SUMMARY:
Phase 2, randomized, open-label study to evaluate the safety and efficacy of maraviroc, favipiravir, and both drugs administered along with currently used therapy in hospitalized patients with pulmonary SARS-CoV-2 (Severe Acute Respiratory Syndrome Coronavirus 2) infection (COVID-19)

DETAILED DESCRIPTION:
The COVID-19 pandemic (Coronavirus Disease-19) caused by SARS-CoV-2 (Severe Acute Respiratory Syndrome Coronavirus 2) has caused more that 10 million infections worldwide, with a general mortality of 6%. Multiple studies have found that the hyperinflammatory immune response induced by SARS-CoV-2 is one of the main causes of severity and death in infected patients. In severe COVID-19 patients, an association was found between pneumonitis and/or ARDS (Acute Severe Respiratory Syndrome), increased serum levels of cytokines and chemokines, extensive lung damage and microthrombosis. Studies of both gene expression in lungs and blood cytokines and chemokines have related chemokine signaling clusters with COVID-19 severity, being CCL3, CCL4 and CCL7 (CC chemokine ligands 3, 4 and 7) particularly interesting. All these are CCR5 (CC chemokine receptor 5) ligands. A strategy to modulate activation and trafficking of leukocytes to the lungs is by blocking CCR5 by using maraviroc (MVC), which has shown capable of modulating conditions of generalized inflammation. Along with a good regulation of the immune response, an antiviral that helps to reduce the viral load must be considered. Favipiravir (FPV) has shown to be capable to reduce the time of viral clearance by half. Hence, we propose that the conjoint use of MVC and FPV could help to reduce the progression of severe hospitalized COVID-19 patients to critical by decreasing the percentage of patients in need of mechanical respiratory support or death by at least 30%. This is a randomized, controlled clinical trial that besides evaluating the safety and efficacy of MVC+FPV to avoid progression in severe COVID-19 patients as a primary endpoint, is also aimed at other secondary endpoints: A) Evaluate the activation of CCR5 in peripheral blood lymphocytes, monocytes, and neutrophils. B) Find possible modifications in the ongoing chemokine and cytokine storm in serum, particularly IL-6, IL-1b, (interleukins 6 and 1 beta) TNF (tumor necrosis factor), IFNa, IFNg (interferons alpha and gamma), VEGF (vascular endothelial growth factor), CXCL10 (CXC chemokine ligand 10), CCL7, CCL3, and CCL5 (CC chemokine ligands 7, 3 and 5), C) Search for alterations in the patterns of activation, trafficking, and exhaustion of peripheral blood lymphocytes, monocytes and neutrophils, and D) Determine if it has an effect in viral loads in saliva. 100 severe patients tested positive for SARS-CoV-2 will be randomized in 4 treatment arms:

Arm A: Currently used therapy (CT) only, Enoxaparin, dexamethasone, and antibiotics if associated bacteremia is present, as per currently used at Hospital General de México "Dr. Eduardo Liceaga").

Arm B: CT+MVC Arm C: CT+FPV Arm D: CT+MVC+FPV

ELIGIBILITY:
Inclusion Criteria:

* With severe non-critical stage of COVID at the time of admission.
* Patients tested positive for SARS-CoV-2 confirmed by PCR (Polymerase Chain Reaction) or quick antigen test
* Within the first 12 days post appearance of symptoms
* With at least one of the following risk factors: Diabetes mellitus (DM), obesity (BMI>30, hypertension, age > 65 years.
* Respiratory rate 25-34/min and no signs of respiratory distress.
* With at least two of the following indicators of severity: SpO2 81-90%, PaFi 150-300 mmHg, FiO2>60% , lung damage in thorax radiographic image => 25% as determined by RALE score (an equivalent to 2-4).
* Normal liver function (Considered up to a fivefold increase above the normal limits of hepatic transaminases)
* Signed informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Patients already participating in another clinical study
* Oxygen saturation < 70% (ambient)
* Clinical evidence of an infectious disease different from COVID at the time of admission
* Chronic kidney failure
* Coronary disease
* Glomerular filtration rate < 30ml/min/1.73 m2 and known history of preexisting chronic renal failure (Chronic kidney disease stages 4-5)
* Known history of HCV, HBV and/or clinical signs of hepatic liver failure.
* Any type of cancer
* HIV and/or any anti retroviral treatment
* Inability to freely decide to participate
* Psychotropics treatment
* Erythromycin treatment
* Polydrug use (Defined as more than two addictions combined)
* With transplant background
* With any autoimmune disorder
* With known hypersensibility to maraviroc and/or favipiravir
* On invasive mechanical ventilation at the time of randomization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Patients free of mechanical ventilation or death | 28 days post start
  Percentage of patients free of mechanical ventilation or death

SECONDARY OUTCOMES:
Patients free of mechanical ventilation or death | 5 days post start
  Percentage of patients free of mechanical ventilation or death
Time of clinical improvement | 15 days post start
  Time of improvement in at least 2 items of the 8-item World Health Organization (WHO) ordinal scale for COVID-19 in days.
Rate of change in phosphorylated CCR5 | Day 10-1
  Rate of change (Delta) in lymphocytes, monocytes and neutrophils with phosphorylated CCR5 as per measured by parameters of flow cytometry.
Rate of change in peripheral blood levels of proinflammatory cytokines and chemokines | Day 10-1
  Rate of change (Delta) in peripheral blood levels of proinflammatory cytokines and chemokines [IL-6, IL-1b, TNF, IFNa, IFNg, VEGF, GM-CSF (granulocyte-macrophage colony stimulating factor), CCL2, CCL3, CCL4, CCL5, CXCL10 and CCL7], as per measured by parameters of flow cytometry
Change in the trafficking and activation pattern of peripheral leukocytes | Day 10-1
  Statistically significant change in the expression of activation [phosphorylated CCR5,CD38, CD126, CD127, CD25, CD86, CD83, CD40 (clusters of differentiation 38, 126, 127, 25, 86 and 40), HLA-DR (Human Leukocyte Antigen-DR isotype), Granzyme B, Perforin, CD107A, CD123, gp130, CD95], trafficking [CCR5, CCR2, CCR6, CCR7, CXCR1, CXCR3 , CXCR5, (CXC chemokine receptors 1, 3 and 5), CX3CR1 (CX3C chemokine receptor] and exhaustion (PD1, programmed death-1 receptor) markers in peripheral blood lymphocytes, neutrophils and monocytes, as per measured by parameters of flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: María Luisa Hernández-Medel, MD, Study Chair — Hospital General de México Dr. Eduardo Liceaga
Locations (1):
- Hospital General de México "Dr. Eduardo Liceaga", Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Inter-institutional exchange of data
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Information will be shared upon completion of the study for collaborative purposes
Access Criteria: Upon request